CLINICAL TRIAL: NCT06006728
Title: Real World Efficacy, Safety of Nanoliposomal Irinotecan With Fluorouracil and Folinic Acid in Metastatic Pancreatic Cancer After Previous Gemcitabine-based Therapy
Acronym: NALIRI-PANC
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/14
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
Keywords: pancreatic adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- naliri: Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy

SUMMARY:
The objectives of the study are to evaluate the efficacy (primary endpoint: overall survival), safety (secondary endpoint) and the medico-economic impact (secondary endpoint) of nanoliposomal irinotecan combined with 5-fluorouracil and folinic acid in clinical practice

DETAILED DESCRIPTION:
Nanoliposomal irinotecan combined with 5-fluorouracil and folinic acid was shown to be effective after gemcitabine-based treatment in patients with metastatic pancreatic adenocarcinoma in the phase III NAPOLI-1 randomized trial.

Nanoliposomal irinotecan is authorized in combination with 5-fluorouracil (5-FU) and leucovorin (LV), as it has shown an improvement in overall survival (median +1.9 months, HR = 0.67) compared to 5-FU/LV alone, without degradation of quality-of-life scales.

However, patients included in clinical trials regularly differ from patients in routine practice, and a real-life study is fundamental in this poor prognosis situation where quality of life preservation is paramount

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* histological or cytological confirmation of pancreatic ductal adenocarcinoma
* measurable lesion(s)
* progression after gemcitabine-based treatment administered in a neoadjuvant, adjuvant protocol (only if remote metastases developed within 6 months of the end of adjuvant treatment), locally advanced, or metastatic phase. They may have already received irinotecan and/or fluorouracil.
* Performance Status (PS) 0 or 1
* Oral consent
* Health insurance

Exclusion Criteria:

* symptomatic brain metastases (cerebral edema, corticosteroids, progressive disease)
* thromboembolic events within six months of inclusion;
* Class III or IV congestive heart failure, ventricular arrhythmia, uncontrolled hypertension.
* Patient under legal protection
* Hypersensitivity to irinotecan
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient treated with nanoliposomal irinotecan with fluorouracil and folinic acid for metastatic pancreatic adenocarcinoma after progression with gemcitabine-based treatment
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 3 years

SECONDARY OUTCOMES:
Response rate to treatment | Every 3 months up to 3 years
  Initial staging at the time of diagnosis is based on computed tomography (CT) or magnetic resonance imaging (MRI).
  Duration of treatment is calculated from the day of nal-IRI initiation to the day of disease progression, switch to other treatment regimens or when the patient is lost to follow-up.
  Tumor response is assessed by abdominal CT or MRI, according to the Response Evaluation Criteria in Solid Tumors (RECIST; version 1.1) and CA19-9.
Progression-free survival | Every 3 months up to 3 years
Cost evaluation | Every 3 months up to 3 years
  number of vials per patient

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No